CLINICAL TRIAL: NCT00003260
Title: Multicentre Phase III Comparing To Therapeutic Sequence: Folfiri Following of Folfox6 (Group A) and Folfox6 Following Of (Group B) For Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Recurrent Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066151; FRE-GERCOR-C97-3/CPTF308; FRE-C97-3/CPTF301; FRE-C97-3/CPTF308; RP-FRE-C97-3/CPTF308; EU-97044
Record Dates: First submitted 1999-11-01; First posted 2004-08-25 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug and giving the drugs in different combinations may kill more tumor cells. It is not yet known whether receiving irinotecan with fluorouracil and leucovorin is more effective than receiving oxaliplatin with fluorouracil and leucovorin in treating recurrent metastatic colorectal cancer

PURPOSE: Randomized phase III trial to compare the effectiveness of irinotecan with oxaliplatin followed by fluorouracil and leucovorin in treating patients with recurrent metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of leucovorin calcium plus fluorouracil with either irinotecan or oxaliplatin in terms of progression free survival in patients with recurrent metastatic colorectal cancer. II. Compare the efficacy, tolerance, quality of life, and overall survival in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by participating institution and measurable or evaluable disease. Patients are randomized to receive either a 2 hour continuous infusion of irinotecan or a 2 hour continuous infusion of oxaliplatin on day 1. All patients receive a 2 hour continuous infusion of leucovorin calcium followed by IV bolus and 48 hour continuous infusion of fluorouracil on days 1 and 2. Courses are repeated every 2 weeks. Patients will receive the alternate treatment if disease progression or unacceptable toxicity occurs on their initial treatment. Patients are followed every 3 months after end of treatment.

PROJECTED ACCRUAL: This study will accrue a total of 109 patients per arm over approximately 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent stage IV adenocarcinoma of the colon and rectum No CNS metastases Bidimensionally measurable lesion (at least 2 cm in dimension) or evaluable disease (as malignant ascites or bone metastases) as documented by CT or MRI Must be outside prior radiotherapy field

PATIENT CHARACTERISTICS: Age: 18 to 75 Performance status: WHO 0-2 Life expectancy: Greater than 3 months Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal Alkaline phosphatase no greater than 3 times normal SGOT/SGPT no greater than 3 times normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No uncontrolled congestive heart failure or angina pectoris in the past 6 months No hypertension or arrhythmia in the past 6 months Neurologic: No peripheral neuropathy No significant neurologic or psychiatric disorder Other: No complete or partial obstruction of the bowel No serious nonmalignant disease No active infection No second malignancy except in situ cervical carcinoma or nonmelanomatous skin carcinoma No chronic diarrhea Not pregnant or nursing Fertile women must use adequate contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior immunotherapy for metastatic disease Chemotherapy: No prior chemotherapy for metastatic disease At least 6 months since prior adjuvant chemotherapy with no disease progression or after metastatic liver resection No prior chemotherapy with oxaliplatin or irinotecan Endocrine therapy: Not specified Radiotherapy: At least 2 weeks since prior radiotherapy Surgery: At least 2 weeks since surgery Other: At least 30 days since use of investigational agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 1998-01

CONTACTS AND LOCATIONS:
Overall Officials: Aimery de Gramont, MD, Study Chair — Hopital Saint Antoine
Locations (1):
- Hopital Saint Antoine, Paris, France